CLINICAL TRIAL: NCT02154672
Title: Prostate Cancer Screening in Men With Germline BRCA2 Mutations
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: 1402013376
Record Dates: First submitted 2014-05-30; First posted 2014-06-03 (Estimated); Results first posted 2021-02-09 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- BRCA2 Carriers: All men identified to have a BRCA2 mutation as part of the Yale Cancer Genetic Counseling Program will be approached and offered participation in the study via our program newsletter, BRCA listserv, Facebook page and a targeted mailing

SUMMARY:
The purpose of this study is to determine the incidence of prostate cancer in men with the BRCa2 gene mutation as an independent indicator for prostate cancer screening.

DETAILED DESCRIPTION:
This is a cohort screening study to prospectively identify the incidence of prostate cancer in a population of BRCA2 carriers. All men identified to have a BRCA2 mutation as part of the Yale Cancer Genetic Counseling Program will be approached and offered participation in the study via our program newsletter, BRCA listserv, Facebook page and a targeted mailing.

Standard of care screening at the Yale Cancer Center for men with a normal prostate cancer risk consists of a PSA test and prostate physical examination beginning at age 50 years and if either is abnormal an MRI of the prostate followed by Fusion-targeted biopsy of the prostate is performed.

ELIGIBILITY:
Inclusion Criteria:

* All men ≥30 years of age with at least a ten-year life expectancy
* A known BRCA2 mutation
* Ability to have an MRI
* Able to give informed consent will be approached to participate in the study

Exclusion Criteria:

* If a man has received or is currently receiving treatment for prostate cancer

Ages: 30 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants will be identified because of their BRCA2 mutation that places them at increased risk for developing prostate cancer. Because this is a pre-selected high-risk population, and our goal is to establish the incidence of cancer and association of risk factors with developing disease, all men ≥30 years of age, able to give informed consent, and with at least a 5-10 year life expectancy will have PSA testing, prostate examination, Pelvic MRI, and Artemis fusion prostate biopsy.
  Men identified to have prostate cancer will be treated according to current standards of care. Treatment for prostate cancer at the Yale Cancer Center is largely based on clinical risk; options include, but are not limited to, active surveillance for appropriate men with low risk disease, treatment with curative intent for men with localized intermediate and high risk prostate cancer, and systemic therapy for men with metastatic disease.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2014-05; Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Preston Sprenkle, MD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BRCA2 Carriers
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | BRCA2 Carriers
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Prostate Cancer Patients With BRCA2 Mutation Carriers
Description: number of patients with a BRCA2 mutation who are diagnosed with prostate cancer
Time Frame: Up to 3 years
Measure: Number; unit: participants
Arm/Group | BRCA2 Carriers
Number analyzed (Participants) | 1
participants | 0

ADVERSE EVENTS:
Time Frame: five years
Arm/Group | BRCA2 Carriers
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-29): https://cdn.clinicaltrials.gov/large-docs/72/NCT02154672/Prot_SAP_000.pdf